CLINICAL TRIAL: NCT06210477
Title: Comparisons of Clinical and Urodynamic Parameters and Persistence in the Treatment for Women With Different Types of Low Bladder Compliance
Brief Title: Association With Low Compliance Bladder in Women With LUTS
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202303086RINC
Record Dates: First submitted 2023-12-22; First posted 2024-01-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Urinary Bladder, Overactive; Urinary Bladder Neck Obstruction; Pelvic Organ Prolapse; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder Neck Obstruction; Pelvic Organ Prolapse; Urinary Incontinence | interventions — Muscarinic Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low compliance: Low urinary tract symptoms with low bladder compliance
  Interventions: Drug: medical treatment for lower urinary tract symptoms

INTERVENTIONS:
Drug: medical treatment for lower urinary tract symptoms — The clinical and urodynamic features on the severity of low compliance bladder in neurologically intact women with lower urinary tract symptoms are indeterminate. Thus, this study aimed to elucidate the above association.
  Other Names: antimuscarinics

SUMMARY:
Hypothesis / aims of study The clinical and urodynamic features on the severity of low compliance bladder in neurologically intact women with lower urinary tract symptoms are indeterminate. Thus, this study aimed to elucidate the above association.

Study design, materials and methods Between January 1996 and December 2021, the medical records of all consecutive women who underwent urodynamic studies for their lower urinary tract symptoms were reviewed to elucidate the clinical significance of low bladder compliance.

ELIGIBILITY:
Inclusion Criteria:

* Urodynamic finding with low bladder compliance

Exclusion Criteria:

* Nil.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women who underwent urodynamic studies
Study Population: Women with lower urinary tract symptoms
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Bladder capacity (mL) | 1996/1/1~2021/12/31
  To compare the bladder capacity (mL) between the groups with and without low bladder compliance. The bladder capacity will be derived from the filling cystometry of urodynamic studies.

SECONDARY OUTCOMES:
Persistence rates of treatment (%) | 1996/1/1~2021/12/31
  To compare the persistence rates of treatment (%) between the groups with and without low bladder compliance. The persistent rate of treatment will be checked from outpatient medical records about prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, MD, PhD, Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital
Locations (1):
- Department of Obstetrics and Gynecology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No